CLINICAL TRIAL: NCT01539460
Title: A Refined Minimally Invasive Procedure for Radical Treatment of Axillary Osmidrosis: Combined Tumescent Liposuction With Subcutaneous Pruning Through a Small Incision
Brief Title: A Minimally Invasive Surgery for Axillary Osmidrosis: Combined Liposuction With Subcutaneous Pruning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, YUEJUN LI, associate professor, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDH0369
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Sweat Gland Diseases
Keywords: Axillary osmidrosis; liposuction; minimally invasive surgery
MeSH Terms: conditions — Sweat Gland Diseases | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- minimally invasive surgery (Experimental): There is only one arm to this study. All patients will receive treatment with the minimally invasive surgery for their axillary bromidrosis
  Interventions: Procedure: minimally invasive surgery

INTERVENTIONS:
Procedure: minimally invasive surgery — Subcutaneous fat and apocrine sweat glands were removed by suction under tumescent anesthesia,and the remaining tissue and glands, tightly attached to the epidermis-dermis interface, were completely removed with scissors through the initial small incision.

SUMMARY:
Patients with axillary osmidrosis are treated with minimally invasive procedure combined tumescent liposuction with Subcutaneous Pruning. Effectiveness of this modified method in reducing odor is to be determined.

DETAILED DESCRIPTION:
Patients with excessive malodor are recruited. They are surgically treated with minimally invasive procedure combined tumescent liposuction with Subcutaneous Pruning and followed up for 6-24 months to evaluate effectiveness sand side effect.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* unpleasant odor from the axillae
* Willing and able to appear for all scheduled, post-operative visits

Exclusion Criteria:

* under the age of 18
* have undergone a prior surgical intervention
* inappropriate candidates for surgery due to medical or mental health reasons
* elect not to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of the refined minimally invasive procedure for radical treatment of axillary osmidrosis using patient self-report assessments | up to 24 months
  the satisfaction of patients

CONTACTS AND LOCATIONS:
Overall Officials: XUEYONG LI, MD, Study Director — Department of Plastics and Burns, Tangdu Hospital
Locations (1):
- Yuejun Li, Xi'an, Shaanxi, China